CLINICAL TRIAL: NCT01802411
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo Controlled Study to Assess the Efficacy and Safety of Intercostal Nerve Block With Liposome Bupivacaine in Subjects Undergoing Posterolateral Thoracotomy
Brief Title: Intercostal Nerve Block With Liposome Bupivacaine in Subjects Undergoing Posterolateral Thoracotomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 402-C-322
Record Dates: First submitted 2013-02-26; First posted 2013-03-01 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Posterolateral Thoracotomy; Postoperative Pain
Keywords: liposome bupivacaine; posterolateral thoracotomy; intercostal nerve block; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EXPAREL 266 mg (Active Comparator): Intercostal nerve block using single total administration of 20 mL EXPAREL (bupivacaine liposome injectable suspension) 266 mg (approximately 88 mg [6.6 mL] to each of three nerve segments)
  Interventions: Drug: EXPAREL 266 mg
- Placebo (Placebo Comparator): Intercostal nerve block using single total administration of 20 mL normal saline (6.6 mL to each of three nerve segments)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EXPAREL 266 mg
  Arms: EXPAREL 266 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to examine the safety and efficacy of liposome bupivacaine for intercostal nerve block in subjects undergoing posterolateral thoracotomy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥18 years of age.
* Scheduled to undergo a thoracotomy of at least 3 inches (7.6 cm) of intercostal incisional length or requiring insertion of an inter-rib spreader/retractor for a primary thoracic non-infectious indication under general anesthesia.
* American Society of Anesthesiologists (ASA) Physical Status 1 - 3.
* Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments.
* Able to demonstrate sensory function by exhibiting sensitivity to cold in one dermatome area in which study drug will be administered.

Exclusion Criteria:

* Currently pregnant, nursing, or planning to become pregnant during the study or within 1 month after study drug administration. Female subjects must be surgically sterile, at least 2 years menopausal, or using an acceptable method of birth control. If of childbearing potential, must have a documented negative pregnancy test within 24 hours before surgery.
* Any planned pleurodesis as part of the surgical procedure.
* Use of any of the following medications within the times specified before surgery: long-acting opioid medication, non-steroidal anti-inflammatory drug (NSAID), or aspirin (except for low-dose aspirin used for cardioprotection or acetaminophen/paracetamol) within 3 days and any opioid medication within 24 hours.
* Use of selective serotonin reuptake inhibitors (SSRIs), gabapentin, pregabalin (Lyrica®), or duloxetine (Cymbalta®) within 3 days of surgery.
* Concurrent painful physical condition or concurrent surgery that may require analgesic treatment (such as an NSAID or opioid) in the postsurgical period for pain that is not strictly related to the surgery, and which may confound the postsurgical assessments (e.g., cancer pain, chronic neuropathic pain, concurrent abdominal surgery).
* Current use of systemic glucocorticosteroids within 1 month of enrollment.
* Body weight < 50 kilograms (110 pounds) or a body mass index ≥ 35 kg/m2.
* Contraindication to any of the pain-control agents planned for surgical or postsurgical use (i.e., fentanyl, morphine, hydromorphone, oxycodone, or bupivacaine).
* Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.
* Previous participation in a liposome bupivacaine study.
* History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
* Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, could interfere with study assessments or compliance.
* Current or historical evidence of any clinically significant disease or condition, especially cardiovascular or neurological conditions that, in the opinion of the Investigator, may increase the risk of surgery or complicate the subject's postsurgical course or interfere with the determination of pain intensity related solely to the surgery.
* Significant medical conditions (including widely disseminated metastatic disease) or laboratory results that, in the opinion of the Investigator, indicate an increased vulnerability to study drugs and procedures.
* Subjects who are planned to receive Entereg® (alvimopan).
* Subjects who will receive prophylactic antiemetics or planned postsurgical antiemetics given without regard to the subject's emesis needs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erol Onel, MD, Study Director — Pacira Pharmaceuticals, Inc
Locations (21):
- United States (7):
  - Jackson Memorial Hospital/University of Miami, 1611 NW 12th Avenue (R-C300), Miami, Florida
  - Louisiana State University Health Sciences Center - Shreveport, 1501 Kings Hwy, Shreveport, Louisiana
  - Sanford Heart Center 801 Broadway North, Fargo, North Dakota
  - Research Concepts, GP, LLC, 4525 Texas St., Bellaire, Texas
  - UT Southwestern Medical Center, Dept. Cardiovas7726cular & Thoracic Surgery, 5909 Harry Hines Blvd., 9th Fl., Dallas, Texas
  - The Methodist Hospital UANEU25, Department of Cardiovascular Surgery, 6550 Fannin, Suite 1401, Houston, Texas
  - MultiCare Health System dba Tacoma General Hospital 315 Martin Luther King Jr Way, Tacoma, Washington
- Bulgaria (4):
  - Thoracic Surgery Clinic, SHATPulmD 'Sveta Sofia', Plovdiv
  - Department of surgery with activity in thoracic surgery, Sofia
  - Military Medical Academy, Sofia
  - University Multiprofile Hospiatl for Active Treatment and Emergency Medicine 'Pirogov', Sofia
- Czechia (3):
  - Krajska nemocnice Liberec, a.s., Vseobecna chirurgie, Liberec
  - Fakultni nemocnice Olomouc I. chirurgicka klinika, Olomouc
  - Thomayerova nemocnice Oddeleni hrudni chirurgie Videnska, Prague
- Georgia (3):
  - Amtel Hospital First Clinical' LLC, Tbilisi
  - Jsc 'National Center for Tuberculosis and Lung Diseases'/, Tbilisi
  - Jsc 'National Center for Tuberculosis and Lung Diseases', Tbilisi
- Poland (4):
  - Klinika Chirurgii Klatki Piersiowej, Chirurgii Ogolnej i Onkologicznej Uniwersytecki Szpital Kliniczny, Lodz
  - Klinika Chirurgii Klatki Piersiowej Pomorskiego Uniwersytetu Medycznego w Szczecinie Specjalistyczny Szpital im. prof. Alfreda Sokolowskiego, Szczecin
  - Oddzial Zabiegowy Kliniki Nowotworow Pluca i Klatki Piersiowej Centrum Onkologii-Instytut im. Marii Sklodowskiej-Curie, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. Prof. Stanislawa Szyszko Slaskiego UM w Katowicach Klinika Anestezjologii i Intensywnej Terapii, Zabrze

RESULTS

PARTICIPANT FLOW:
Groups:
- EXPAREL 266 mg: Intercostal nerve block using single total administration of 20 mL EXPAREL (bupivacaine liposome injectable suspension) 266 mg (approximately 88 mg [6.6 mL] to each of three nerve segments)
  EXPAREL 266 mg
- Placebo: Intercostal nerve block using single total administration of 20 mL normal saline (6.6 mL to each of three nerve segments)
  Placebo
Period: Overall Study
Arm/Group | EXPAREL 266 mg | Placebo
Started | 96 | 95
Completed | 82 | 74
Not Completed | 14 | 21
Not completed — Death | 2 | 1
Not completed — Adverse Event | 2 | 7
Not completed — Lack of Efficacy | 8 | 10
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Planned pleurodesis as part of the proc | 1 | 0
Not completed — Surgery aborted after bronchoscopy | 1 | 0
Not completed — Proc changed to video-asst thorascopic | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were analyzed in the safety population, which included all participants who received study drug, with analysis based on actual treatment received. Six randomized participants (2 in the EXPAREL 266 mg group and 4 in the placebo group) did not receive study drug and were excluded from the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | EXPAREL 266 mg | Placebo | Total
Number analyzed (Participants) | 94 | 91 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (12.71) | 58.5 (13.03) | 58.2 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 61
  Male | 64 | 60 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 90 | 88 | 178
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 94 | 91 | 185
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5
  Poland | 38 | 32 | 70
  Bulgaria | 20 | 28 | 48
  Czechia | 17 | 18 | 35
  Georgia | 17 | 10 | 27
American Society of Anesthesiologists (ASA) classification [Count of Participants; unit: Participants] — American Society of Anesthesiologists (ASA) classification was determined by physicians using the ASA Physical Status Classification System which assesses the patient's pre-anesthesia medical co-morbidities. ASA 1 patients would be considered a normal, healthy patient. ASA 2 is a patient with mild systemic disease (eg, smoker, well controlled diabetes or high blood pressure (HBP)). ASA 3 is a patient with severe systemic disease (eg poorly controlled diabetes or HBP). ASA 4 is a patient with severe systemic disease that is a constant threat to life (eg, recent myocardial infarction, stroke).
  Participants
    1 | 32 | 24 | 56
    2 | 48 | 50 | 98
    3 | 14 | 17 | 31

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) of Pain Intensity at Rest Through 72 Hours
Description: AUC of pain intensity scores at rest through 72 hours postsurgery. Participants assumed a resting position that did not exacerbate his or her postsurgical pain. Pain intensity scores were measured at baseline and 1, 2, 4, 8, 12, 24, 36, 48, 60, and 72 hours postsurgery, at first request for rescue pain medication, and on day 12 using the numeric rating scale at rest (NRS-R; 0=no pain and 10=worst possible pain).
Time Frame: 0-72 hours postsurgery
Population: The efficacy population included all participants who received study drug, with analysis based on randomized treatment
Measure: Least Squares Mean (Standard Error); unit: score on a scale * hr
Arm/Group | EXPAREL 266 mg | Placebo
Number analyzed (Participants) | 94 | 91
score on a scale * hr | 472.1 (37.19) | 459.0 (36.57)
Statistical Analysis 1: Comparison: EXPAREL 266 mg vs Placebo; Test type: Superiority; p = 0.5598, ANCOVA; LSMD = 13.1, 95% CI 2-sided [-31 to 57]

2. Secondary Outcome: Total Postsurgical Opioid Consumption Through 72 Hours
Description: Total postsurgical opioid consumption (morphine equivalent) through 72 hours postsurgery
Time Frame: 0-72 hours postsurgery
Population: The efficacy population included all participants who received study drug, with analysis based on randomized treatment
Measure: Mean (Standard Deviation); unit: mg morphine equivalent dose
Arm/Group | EXPAREL 266 mg | Placebo
Number analyzed (Participants) | 94 | 91
mg morphine equivalent dose | 70.88 (37.537) | 71.38 (39.418)

3. Secondary Outcome: Time to First Opioid Rescue Through 72 Hours Postsurgery
Description: Time to first use of opioid rescue medication through 72 hours postsurgery, calculated as the date and time of first opioid use minus the date and time of the end of surgery.
Time Frame: 72 hours postsurgery
Population: Time to first use of opioid rescue medication through 72 hours postsurgery, calculated as the date and time of first opioid use minus the date and time of the end of surgery.
Measure: Median (Full Range); unit: hours
Arm/Group | EXPAREL 266 mg | Placebo
Number analyzed (Participants) | 94 | 91
hours | 1.1 [0.08 to 72.00] | 0.7 [0.10 to 72.00]

ADVERSE EVENTS:
Time Frame: From time of randomization through the day 30 follow-up contact
Description: The safety population included all participants who received study drug, with analysis based on actual treatment received. Treatment-emergent adverse events that were solicited from the neurological assessment or from the opioid-related AE questionnaire were included in this table.
Arm/Group | EXPAREL 266 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 2/94 | 4/91
Serious Adverse Events (participants affected / at risk) | 12/94 | 10/91
Other Adverse Events (participants affected / at risk) | 63/94 | 55/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EXPAREL 266 mg (N=94) | Placebo (N=91)
Cardiac Arrest (Cardiac disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Lung infection Pseudomonal (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Postprocedural hemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Heart injury (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Acute renal failure (Renal and urinary disorders) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Cerebral hematoma (Nervous system disorders) | 0 | 1
Coma uremic (Nervous system disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EXPAREL 266 mg (N=94) | Placebo (N=91)
Atrial fibrillation (Cardiac disorders) | 2 | 6
Pyrexia (General disorders) | 16 | 12
Hypertension (Vascular disorders) | 10 | 5
Hypotension (Vascular disorders) | 2 | 6
Nausea (Gastrointestinal disorders) | 9 | 7
Vomiting (Gastrointestinal disorders) | 9 | 8
Constipation (Gastrointestinal disorders) | 7 | 4
Fatigue (General disorders) | 9 | 4
Confusional state (Psychiatric disorders) | 7 | 4
Dysgeusia (Nervous system disorders) | 7 | 2
Pruritus generalized (Skin and subcutaneous tissue disorders) | 2 | 5

LIMITATIONS AND CAVEATS:
Study drug delivery to the intercostal nerve via instillation, not US-guided injection, likely prevented optimal placement/retention, as supported by pharmacokinetic data. Thus, efficacy of study drug as regional nerve block could not be meaningfully evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any proposed publication/presentation of study-related information is subject to advance review by the Sponsor ≥60 days before intended submission/presentation. Investigator/institution shall amend publication/presentation as needed to address errors or confidential information identified by the Sponsor. If requested in writing by the Sponsor, investigator/institution shall withhold publication for an additional 90 days.

DOCUMENTS (2):
  • Study Protocol (2012-09-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT01802411/Prot_000.pdf
  • Statistical Analysis Plan (2013-02-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT01802411/SAP_001.pdf